CLINICAL TRIAL: NCT05982587
Title: PanCareSurPass (PCSP) Conduct and Analysis of the Multi-country Implementation Study of the SurPass v2.0
Brief Title: PCSP Implementation Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Riccardo Haupt, Principal investigator, Istituto Giannina Gaslini
Other Study IDs: N.CET-Liguria:265-2023-DB13200
Record Dates: First submitted 2023-07-28; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Survivorship; Late Effect
MeSH Terms: interventions — Calcium Carbonate; Parturition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survivorship passport (SurPass) delivery — The Survivorship Passport (SurPass) is a digital tool developed thanks to several EU projects to help Childhood Cancer Survivors (CCS), their families and health care providers (HCPs) in the follow-up process after completion of anticancer treatment. It comprises two main components: Treatment Summary including demographic, diagnosis and treatment data and personalized Survivorship Care Plan providing individual follow-up care recommendations The SurPass assists both CCS and HCPs to improve Long-Term Follow-Up care, in a partnership, supporting CCS empowerment and satisfaction with care, as well as shared decision-making by CCS and HCPs.
  The aim of the PCSP implementation study is to evaluate feasibility and outcomes (personal and economic) of implementing the SurPass v2.0 in six clinics located in Austria, Belgium, Germany, Italy, Lithuania and Spain by using interoperability procedures according to Health Level 7- Fast Healthcare Interoperability Resource (HL7-FHIR) standards.

SUMMARY:
This study protocol describes the design and methods of the PanCareSurPass (PCSP) multi-country implementation study of the Survivorship Passport v2.0 (short: PCSP implementation study), which is part of the PCSP project that has received funding through the European Union (EU) Horizon 2020 Programme. The cohort study will inform researchers and stakeholders on the process and outcomes of implementing the Survivorship Passport (SurPass) v2.0 in the Electronic Health Information Systems (EHIS) of six clinics in the EU countries Austria (CCRI), Belgium (KU Leuven), Germany (UMC-Mainz/UzL), Italy (IGG), Lithuania (VULSK) and Spain (HULAFE).

The SurPass comprises two main components, the Treatment Summary (TS) including demographic, diagnosis and treatment data and the personalized Survivorship Care Plan (SCP) including individual follow-up care recommendations. The SCP is based on internationally approved, organ-specific follow-up care recommendations.

The SurPass is used as a tool to assist both Childhood Cancer Survivors (CCS) and Health Care Providers (HCPs) to improve Long-Term Follow-Up (LTFU) care, in a care partnership, supporting CCS empowerment and satisfaction with care, as well as shared decision-making by CCS and HCPs. People-centred care is important in CCS since they are a vulnerable population known to be at higher risk of developing chronic conditions as compared to their peers in the general population.

The overall aim of the cohort study is to evaluate the implementation of the SurPass v2.0 in the six centres by testing the feasibility of test wise implementation of the SurPass v2.0 in different health system scenarios and assessing the people-centred LTFU care for CCS with the SurPass as a tool and the cost effectiveness. Six long term follow-up clinics across Europe will enrol eligible, consented CCS and generate personalised digital SurPass. Eligible participants for the main study cohort will be CCS more than 5 years after diagnosis and with an identified treatment burden based on actual exposure to respective treatments (Cumulative Treatment Doses (CTD) of chemotherapy, immunotherapy, radiotherapy). In preparation of the clinic visit, HCPs/local data monitors will use the SurPass v2.0 platform to generate the TS (semi-automated or manual data entry) from which, in turn, the preliminary SCP is automatically created using the built-in algorithms for each consented survivor.

During the clinic visit the preliminary SCP is discussed with the Survivor, and tailored to meet the CCS personal needs and a final SCP will be generated. The SCP will include detailed country-specific recommendations, where applicable. The SurPass v2.0 (TS + SCP) will then be integrated into the institutional EHIS, as well as in the survivor's national/regional Electronic Health Platform (EHP) where available.

CCS who give informed consent will complete (online) study questionnaires at two measuring points: before the visit to the clinic, and after they received the SurPass during the clinical visit. HCPs will also provide study data: the TS which went into the SurPass (clinical data) and data to monitor the implementation and assess the barriers and facilitators of implementing the SurPass. In addition, data will be collected from both survivors and health care providers to assess the cost-effectiveness of implementing the SurPass.

Regarding the outcome evaluation, the main outcome is the change in levels of activation of survivor or caregiver, as assessed using the Patient Activation Measure (PAM) prior and after clinic visit. Further measurements will be made related to: empowerment, satisfaction with the digital SurPass tool, emotional impacts, quality of life and additional costs of CCS.

The main outcome will be analysed by multivariable logistic regression. Analysis for the secondary outcomes will be mostly descriptive. The economic assessment will be analysed by cost analysis, cost utility analysis and multi-criteria decision analysis.

The study will be conducted in accordance with the guidelines of good clinical practice (ICH/GCP) and the Helsinki Declaration. The investigators will carefully address all ethical, legal and safety aspects of the study and fully comply with prevailing national and EU regulations and legislation.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with cancer before the age of 18 years;
* have completed the planned treatment protocol;
* being still in continuous, complete remission at least five years from primary cancer diagnosis (≥5 years survivorship);
* being in follow-up care at one of the institutions participating in the study;
* have signed informed consent/assent to the study according to local legislation.

Exclusion Criteria:

* currently in treatment for secondary malignancy or relapse of primary malignancy;
* have already received previous versions of the SurPass (v1.0 - 1.2).

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Within this study we'll enroll childhood cancer survivors (CCS), defined as those subjects who have survived ≥5 years since diagnosis.
  Compared to the general population, CCS represent a vulnerable population being at increased risk of developing psychosocial and health problems known as late effects, resulting in low quality of life, excess morbidity and mortality
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Study of activation after the delivery of the personal SurPass v2.0 | Before (2-8 weeks) and after (2-3 months) SurPass delivery
  The change in levels of activation after the delivery of the personal SurPass v2.0. Activation will be measured using the validated Patient Activation Measure (PAM). This instrument is a Likert type questionnaire in which respondent score each item with their level of agreement ranging from 1 (strongly disagree) to 4 (strongly agree). In case of the item is not applicable, no score is provided and marked in a specific section.

SECONDARY OUTCOMES:
Study of empowerment after the delivery of the personal SurPass v2.0 | Before (2-8 weeks) and after (2-3 months) SurPass delivery
  The change in levels of empowerment after the delivery of their personal SurPass v2.0. Empowerment will be measured using the validated Health Education Impact Questionnaire (heiQ) scale. This instrument is a Likert type questionnaire in which respondent score each item with their level of agreement ranging from 1 (strongly disagree) to 4 (strongly agree).
Study of CCS quality of life | Before (2-8 weeks) and after (2-3 months) SurPass delivery
  CCS quality of life will be measured using the EuroQoL-5 Dimension (EQ-5D) questionnaire. This instrument is a Likert type questionnaire in which respondent score each quality of life related item ranging from 1 (I have no problems) to 5 (I have major problems).
Study of satisfaction of HCPs and CCS with the digital SurPass tool | At SurPass delivery and after (2-3 months)
  Satisfaction of HCPs and CCS with the digital SurPass tool (either incorporated in the institutional EHIS and/or in national/regional EHP (where available) will be assessed using the validated Technology Acceptance Model (TAM) scale.
  This instrument is a Likert type questionnaire in which respondent score each item with their level of agreement ranging from 1 (strongly agree) to 7 (strongly disagree).
Study of emotional impact after the delivery of the personal SurPass v2.0 | After (2-3 months) SurPass delivery
  The emotional impact of the SurPass delivery on CCS daily life in terms of modifications in daily activities, anxiety related to possible late effects, change in quantity and quality of information regarding possible late effects. This outcome will be evaluated by means of an ad hoc Likert-type PanCareSurPass specific questionnaire (PCSP-Q).
  This instrument is a Likert type questionnaire in which respondent score each item with their level of agreement ranging from 1 (strongly disagree) to 4 (strongly agree). In case of not willing to respond to the specific item, no score is provided and marked in a specific section.
Study of economical impact after the delivery of the personal SurPass v2.0 | Imp-Cost questionnaire: baseline at SurPass delivery. Op-Cost: immediately after SurPass delivery. CCS Cost Qx: within 3 months after SurPass delivery.
  Three different types of costs: (1) costs related to technological development, implementation of interfaces, process adaptations, and social innovation (Imp-Cost), (2) operational costs incurred by the health care providers (Op-Cost) and (3) additional costs of CCS (or their caregivers) regarding the clinical visit (CCS Cost Qx) will be measured using PanCareSurPass specific questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Giannina Gaslini, Genoa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haupt R, Spinetta JJ, Ban I, Barr RD, Beck JD, Byrne J, Calaminus G, Coenen E, Chesler M, D'Angio GJ, Eiser C, Feldges A, Gibson F, Lackner H, Masera G, Massimo L, Magyarosy E, Otten J, Reaman G, Valsecchi MG, Veerman AJ, Penn A, Thorvildsen A, van den Bos C, Jankovic M; International Berlin-Frankfurt-Munster Study Group Early and Late Toxicity Educational Committee (I-BFM-SG ELTEC). Long term survivors of childhood cancer: cure and care. The Erice statement. Eur J Cancer. 2007 Aug;43(12):1778-80. doi: 10.1016/j.ejca.2007.04.015. Epub 2007 May 31. PMID 17543517
- [Background] Jankovic M, Haupt R, Spinetta JJ, Beck JD, Byrne J, Calaminus G, Lackner H, Biondi A, Oeffinger K, Hudson M, Skinner R, Reaman G, van der Pal H, Kremer L, den Hartogh J, Michel G, Frey E, Bardi E, Hawkins M, Rizvi K, Terenziani M, Valsecchi MG, Bode G, Jenney M, de Vathaire F, Garwicz S, Levitt GA, Grabow D, Kuehni CE, Schrappe M, Hjorth L; participants in PanCare. Long-term survivors of childhood cancer: cure and care-the Erice Statement (2006) revised after 10 years (2016). J Cancer Surviv. 2018 Oct;12(5):647-650. doi: 10.1007/s11764-018-0701-0. Epub 2018 Jun 26. PMID 29946794
- [Background] Haupt R, Essiaf S, Dellacasa C, Ronckers CM, Caruso S, Sugden E, Zadravec Zaletel L, Muraca M, Morsellino V, Kienesberger A, Blondeel A, Saraceno D, Ortali M, Kremer LCM, Skinner R, Roganovic J, Bagnasco F, Levitt GA, De Rosa M, Schrappe M, Hjorth L, Ladenstein R; PanCareSurFup, ENCCA Working Group; ExPo-r-Net Working Group. The 'Survivorship Passport' for childhood cancer survivors. Eur J Cancer. 2018 Oct;102:69-81. doi: 10.1016/j.ejca.2018.07.006. Epub 2018 Aug 20. PMID 30138773
- [Background] van Kalsbeek RJ, Mulder RL, Haupt R, Muraca M, Hjorth L, Follin C, Kepak T, Kepakova K, Uyttebroeck A, Mangelschots M, Winther JF, Loonen JJ, Michel G, Bardi E, Elmerdahl Frederiksen L, den Hartogh J, Mader L, Roser K, Schneider C, Brown MC, Brunhofer M, Gottgens I, Hermens RPMG, Kienesberger A, Korevaar JC, Skinner R, van der Pal HJH, Kremer LCM. The PanCareFollowUp Care Intervention: A European harmonised approach to person-centred guideline-based survivorship care after childhood, adolescent and young adult cancer. Eur J Cancer. 2022 Feb;162:34-44. doi: 10.1016/j.ejca.2021.10.035. Epub 2021 Dec 22. PMID 34953441
- [Background] van Kalsbeek RJ, van der Pal HJH, Kremer LCM, Bardi E, Brown MC, Effeney R, Winther JF, Follin C, den Hartogh J, Haupt R, Hjorth L, Kepak T, Kepakova K, Levitt G, Loonen JJ, Mangelschots M, Muraca M, Renard M, Sabic H, Schneider CU, Uyttebroeck A, Skinner R, Mulder RL. European PanCareFollowUp Recommendations for surveillance of late effects of childhood, adolescent, and young adult cancer. Eur J Cancer. 2021 Sep;154:316-328. doi: 10.1016/j.ejca.2021.06.004. Epub 2021 Jul 29. PMID 34333209